CLINICAL TRIAL: NCT07383168
Title: The Effect of Preoperative Education Delivered Using the Pecha Kucha Method on the Quality of Recovery in Individuals Undergoing Cataract Surgery: A Randomized Controlled Study
Brief Title: The Effect of Preoperative Education Delivered Using the Pecha Kucha Method on the Quality of Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09.04.2025/12
Record Dates: First submitted 2026-01-22; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Cataract; Education of Patients; Postoperative Recovery
MeSH Terms: conditions — Cataract | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: After obtaining the necessary approvals, participants were randomly assigned to either the intervention group (n = 31) or the control group (n = 30) using randomization. On the morning of surgery, both groups completed the sociodemographic data form and the QoR-15 questionnaire through face-to-face interviews conducted by the researchers. Following data collection, patients in the intervention group received preoperative education using the Pecha Kucha technique. This education consisted of a 6-minute and 40-second presentation delivered via a smartphone, comprising 20 slides with intensive visual content and minimal text.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): After obtaining the necessary approvals, participants were randomly assigned to either the intervention group or the control group using randomization. On the morning of surgery, both groups completed the sociodemographic data form and the QoR-15 questionnaire through face-to-face interviews conducted by the researchers.
- Study Group (Experimental): After obtaining the necessary approvals, participants were randomly assigned to either the intervention group (n = 31) or the control group (n = 30) using randomization. On the morning of surgery, both groups completed the sociodemographic data form and the QoR-15 questionnaire through face-to-face interviews conducted by the researchers. Following data collection, patients in the intervention group received preoperative education using the Pecha Kucha technique. This education consisted of a 6-minute and 40-second presentation delivered via a smartphone, comprising 20 slides with intensive visual content and minimal text
  Interventions: Other: Education with Pecha Kucha

INTERVENTIONS:
Other: Education with Pecha Kucha — After obtaining the necessary approvals, participants were randomly assigned to either the intervention group (n = 31) or the control group (n = 30) using randomization. On the morning of surgery, both groups completed the sociodemographic data form and the QoR-15 questionnaire through face-to-face interviews conducted by the researchers. Following data collection, patients in the intervention group received preoperative education using the Pecha Kucha technique. This education consisted of a 6-minute and 40-second presentation delivered via a smartphone, comprising 20 slides with intensive visual content and minimal text.
  Arms: Study Group

SUMMARY:
Objective: The aim of this research is to determine the effect of the Pecha Kucha training method on the quality of patient recovery in patient education.

Methods: This study was conducted at the ophthalmology clinic of a training and research hospital in Türkiye. A total of 61 patients scheduled for cataract surgery were randomly assigned to either the intervention group (n = 31) or the control group (n = 30). The study group received preoperative education using the Pecha Kucha method. Data were collected face-to-face using a sociodemographic data form and the Quality of Healing-15 (QoR-15) questionnaire. Data were analyzed using descriptive statistics and appropriate parametric and non-parametric tests, with a statistical significance level of p < 0.05.

DETAILED DESCRIPTION:
this study was conducted to determine the effect of preoperative education delivered using the Pecha Kucha method on recovery in patients undergoing cataract surgery. Additionally, the study aims to highlight the importance of using alternative educational methods to enhance the effectiveness of preoperative education.

ELIGIBILITY:
Inclusion Criteria:

The study sample consisted of patients who agreed to participate and were scheduled for cataract surgery

Exclusion Criteria:

Exclusion criteria included being under 18 years of age and having cognitive impairments that would prevent participation in educational activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2026-01-02 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery-15 (QoR-15) | the morning of the surgery day, 24 hours after the surgery
  The original scale was developed by Myles et al. (2000) to assess postoperative recovery quality¹⁷, and a shortened 15-item version was later developed by Stark et al.¹⁸. The Turkish validity and reliability study was conducted by Kara et al. in 2022. The scale consists of five subdimensions: pain, physical comfort, physical independence, psychological support, and emotional state. Each item is scored on a scale from 0 to 10, with total scores ranging from 0 to 150. Scores between 136-150 indicate excellent recovery, 122-135 good recovery, 90-121 moderate recovery, and 0-89 poor recovery¹⁹.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want to share it until it's published.